CLINICAL TRIAL: NCT01126892
Title: An Open-label, Multicenter Study of Treatment With Nilotinib in Adult Patients With Imatinib - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Brief Title: A Study of Nilotinib in Adult Patients With Imatinib Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Acronym: ENACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ACO01
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Advanced Disease,; Resistance,; Intolerance
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
A multicenter, open label study of Nilotinib in CML patients PH + with imatininb resistant in blast crisis, accelerated phase or chronic phase. The main purpose is evaluate the safety and efficacy of Nilotinib.

ELIGIBILITY:
Inclusion Criteria:

Stratum 1:

1. Currently participating in Novartis study CAMN107A2109
2. Written signed and dated informed consent prior to any study procedures being performed

Stratum 2:

1. Male or female
2. > 18 years
3. ECOG 0,1,2
4. ASL/ALT <= 2.5 ULN or <= 5.0 ULN
5. Alcaline Phosfatase <= 2.5 ULN
6. Serum Bilirrubin <= 1.5 ULN
7. Serum Creatinine <= 1.5 ULN or creatinine clearance >=50 ml/min / 24 hours
8. Serum Lipase <= 1.5 ULN

Exclusion Criteria:

Stratum 1 and stratum 2:

1. Reduction of the cardiac function
2. Use of Coumadin
3. Other severe medical concurrent conditions
4. Treatment with medications that prolonged the QT interval.
5. Mayor surgery 15 days before the inclusion in the protocol
6. Pregnant women or lactation

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maintain and monitor long-term hematological and cytogenetic responses previously obtained by patients participating in the CAMN107A2109 study. | between 6 and 12 months

SECONDARY OUTCOMES:
To evaluate the rate of any durable cytogenetic response and Complete cytogenetic response | 24 months
To evaluate the rate of molecular response every 3 months, until 24th month of treatment or end of study | 24 months
To follow loss of HR (after previous confirmed HR for AP and CHR for CP) | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (2):
- Hospital San José, Bogotá, Colombia, Bogotá, Colombia
- Banco Municipal de Sangre, Caracas, Venezuela